CLINICAL TRIAL: NCT02628925
Title: Nu-DESC DK: The Danish Version of the Nursing Delirium Screening Scale (Nu-DESC DK)
Brief Title: Nu-DESC DK: The Danish Version of the Nursing Delirium Screening Scale
Acronym: Nu-DESC DK
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DHAG-001-2014
Record Dates: First submitted 2015-11-27; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Delirium
Keywords: mass screening; Nursing diagnosis; Psychiatric Status Rating Scale
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Recovery room: 10 medical staff working in the recovery room
  Interventions: Device: Nu-DESC DK
- Orthopedic ward: 10 medical staff working on the orthopedic ward
  Interventions: Device: Nu-DESC DK

INTERVENTIONS:
Device: Nu-DESC DK — Nu-DESC DK as a screening tool is presented to the medical staff and they have to evaluate the tool an evaluate the screening tool on a evaluation form and rates on a 6 step Likert scale.

SUMMARY:
Delirium is one of the most common complications among elderly hospitalized patients, postoperative patients and patients on intensive care units. The reported prevalence is between 11 and 80 %. Delirium is associated with a high morbidity and threefold higher 6-month mortality. The Nursing-Delirium Screening Scale (Nu-DESC) is a screening tool with a high sensitivity and specificity.

The purpose of this study is to translate the Nu-DESC to danish and evaluate afterwards its feasibility and understanding by different medical staff.

Material and methods:

The Nu-DESC will be translated after International Society for Pharmacoeconomics and Outcomes Research (ISPOR) guidelines to Danish by permission of the original author.

The evaluation will be performed, by filling out evaluation forms, where the feasibility and understanding will be rated on a 6 step Likert scale.

DETAILED DESCRIPTION:
Translation of the original tool and evaluation of understanding and feasibility by medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Medical staff working in the recovery room or orthopedic ward

Exclusion Criteria:

* Medical staff from other wards

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical staff on 2 different wards
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference in understanding of the content of Nu-DESC DK by different medical staff groups | Within the first week after questionnaire is filled out
  All five sections of Nu-DESC DK will each be rated on a 6 step Likert scale regarding language and content.
Difference in feasibility of the content of Nu-DESC DK by different medical staff groups | Within the first week after questionnaire is filled out
  All five sections of Nu-DESC DK will each be rated on a 6 step Likert scale regarding time and usability